CLINICAL TRIAL: NCT02144558
Title: Evolution of Sperm Parameters and Study of Risk Factors of Impairment of Sperm Quality in Spinal Cord Injuries. Longitudinal Prospective Study.
Brief Title: Fertility of Spinal Cord Injured Men
Acronym: FertiSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence de La Biomédecine (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P130703
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sperm Parameters of Spinal Cord Injured Men
Keywords: Sperm parameters; Spinal cord injuries; Oxidative stress; Inflammatory syndrome
MeSH Terms: conditions — Spinal Cord Injuries | interventions — poliovirus receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal cord injured (SCI) men, para or tetraplegic (Experimental): SCI men will have 4 medical visits associated to sperm retrieval (penile vibratory stimulation (PVS) or masturbation)
  Interventions: Other: penile vibratory stimulation (PVS) or masturbation

INTERVENTIONS:
Other: penile vibratory stimulation (PVS) or masturbation — penile vibratory stimulation (PVS) or masturbation

SUMMARY:
Spinal cord injured (SCI) men, para or tetraplegic, most often have an infertility, caused among others by a deficiency of sperm quality particularly motility and vitality. Several mechanisms have been proposed: low frequency of ejaculation, recurrent urinary tract and seminal infections, presence of an inflammatory syndrome (IS) and an oxidative stress (OS). However, no French study of sperm quality has been conducted in this population that could identify aggravating factors of sperm quality and a way to prevent them.

Hypothesis: Sperm parameters decrease rapidly following spinal cord injury and next stabilise. However, unidentified yet risk factors could influence long-term evolution of sperm parameters.

The objective is to study the evolution of sperm parameters during 18 months taking into account bladder management, recurrent urinary tract and bladder infections, IS and OS. The evaluation of these parameters and their consequences will be indicative to determine one or more risk factors of sperm degradation and determine a strategy for long term support to avoid the use of ART either by sperm cryopreservation and/or by preventing risk factors

DETAILED DESCRIPTION:
SCI men are mostly young adults who have not completed their parental project. Infertility has many causes: erectile dysfunction, anejaculation (85% of SCI ) and altered sperm parameters. Penile vibratory stimulation allows 75 % of the sperm collection. If sperm quality is sufficient, intravaginal insemination of their partner at home is possible. The use of AMP remains common, which is damaging to men non sterile priori. In SCI, sperm concentration remains satisfactory but mobility and vitality are impaired. The installation of this irreversible degradation likely occurs very quickly after the trauma. The possible deterioration of sperm parameters with time is not known. The following pathophysiological mechanisms have been proposed: i) increased scrotal temperature, ii) decreased ejaculatory frequency, iii) recurrent urinary tract and seminal infections, iv ) inflammation and oxidative stress in the semen. Patients, and even rehabilitation doctors often submit an application for preventive sperm conservation but in the absence of prospective longitudinal data on the evolution of sperm quality of SCI men over the time and identified risk factors of degradation, the indication and timing of preventive cryopreservation remain to be defined.

Hypothesis: The sperm parameters, mobility and vitality, in SCI patients with or without penile vibratory stimulation (PVS), decrease in the immediate aftermath of trauma and next stabilize out the occurrence of intercurrent medical events or symptomatic urogenital infections. However, unidentified yet risk factors could influence long-term evolution of these sperm parameters.

Main objective: Monitoring the evolution of sperm parameters for 18 months: concentration, mobility, vitality, sperm morphology, inflammatory syndrome and oxidative stress on 4 ejaculates collected by masturbation or SVP at 6-month intervals.

Secondary objectives: In case of impaired sperm quality, identify risk factors for this change.

SCI men will have 4 medical visits associated to sperm retrieval spaced to 6 months during 18 months. At each visit medical and reproductive informations will be collected.

Knowledge of the evolution of sperm parameters and risk factors of its degradation over time must answer with the criteria of "evidence based medicine" the request of sperm cryopreservation frequently expressed by SCI patients. This study should lead to the optimization of the management of infertility in patients with spinal cord injuries and giving directions for research aiming to prevent the degradation of sperm parameters. Finally, this study should provide the rationale for future research on clinical risk factors and / or biological degradation of sperm and biological markers of risk of degradation.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injured men aged between 18 and 60 years
* Strict antegrade ejaculation obtained by masturbation or penil vibratory stimulation
* Signature of an informed and written consent to participate to the study.

Exclusion Criteria:

* Total or partial retrograde ejaculation
* Major patients protected
* Men no affiliated with a french social security regime.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Sperm viability: percent of live spermatozoa among 100 counted spermatozoa. | 18 month
  Sperm viability is a stable criteria of evaluation and it has a good repeatability in our lab.
  Sperm viability is measured on fresh sperm 30 minutes after ejaculation using eosine nigrosine coloration. This measure is repeated on each of the four ejaculates obtained at 6 months apart.

SECONDARY OUTCOMES:
spermogram | 18 months
  Sperm concentration, mobility and morphology
elastase | 6 month
  Measure of inflammation
DNA fragmentation | 18 months
  Sperm DNA integrity, measures oxidative stress
8 Hydroxydesoxyguanosine (8OHdG) | 18 months
  Oxydative stress
Seminal biochemistry | 18 months
  Secretion of seminal tract
Urinary and seminal infections | 18 months
  Bacteriological analysis of sperm and urine
Mode of urinary catheter | 18 months
Spinal cord injury type | 0 months
  Type and level of the lesion
Concomitant treatments | 18 months
Patient age and time to spinal cord injury | 18 months
Sperm viability: percent of live spermatozoa among 100 counted spermatozoa. | 6 months
  Sperm viability is a stable criteria of evaluation and it has a good repeatability in our lab.
  Sperm viability is measured on fresh sperm 30 minutes after ejaculation using eosine nigrosine coloration. This measure is repeated on each of the four ejaculates obtained at 6 months apart.
Sperm viability: percent of live spermatozoa among 100 counted spermatozoa. | 12 months
  Sperm viability is a stable criteria of evaluation and it has a good repeatability in our lab.
  Sperm viability is measured on fresh sperm 30 minutes after ejaculation using eosine nigrosine coloration. This measure is repeated on each of the four ejaculates obtained at 6 months apart.
Sperm viability: percent of live spermatozoa among 100 counted spermatozoa. | 0 months
  Sperm viability is a stable criteria of evaluation and it has a good repeatability in our lab.
  Sperm viability is measured on fresh sperm 30 minutes after ejaculation using eosine nigrosine coloration. This measure is repeated on each of the four ejaculates obtained at 6 months apart.
elastase | 0 month
  Measure of inflammation
elastase | 12 month
  Measure of inflammation
elastase | 18 month
  Measure of inflammation
spermogram | 0 months
  Sperm concentration, mobility and morphology
spermogram | 6 months
  Sperm concentration, mobility and morphology
spermogram | 12 months
  Sperm concentration, mobility and morphology
DNA fragmentation | 0 month
  Sperm DNA integrity, measures oxidative stress
DNA fragmentation | 6 months
  Sperm DNA integrity, measures oxidative stress
DNA fragmentation | 12 months
  Sperm DNA integrity, measures oxidative stress
8 Hydroxydesoxyguanosine (8OHdG) | 0 months
  Oxydative stress
8 Hydroxydesoxyguanosine (8OHdG) | 6 months
  Oxydative stress
Seminal biochemistry | 0 months
  Secretion of seminal tract
Seminal biochemistry | 6 months
  Secretion of seminal tract
Seminal biochemistry | 12 months
  Secretion of seminal tract
Urinary and seminal infections | 0 months
  Bacteriological analysis of sperm and urine
Urinary and seminal infections | 6 months
  Bacteriological analysis of sperm and urine
Urinary and seminal infections | 12 months
  Bacteriological analysis of sperm and urine
Mode of urinary catheter | 0 months
Mode of urinary catheter | 6 months
Mode of urinary catheter | 12 months
Concomitant treatments | 0 month
Concomitant treatments | 6 months
Concomitant treatments | 12 months
Patient age and time to spinal cord injury | 0 month
Patient age and time to spinal cord injury | 6 months
Patient age and time to spinal cord injury | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Céline Chalas, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Assistance Publique-Hôpitaux de Paris, Cochin Hospital, Department of Biology of Reproduction, Paris, France

REFERENCES:
- [Background] Chalas C, Jilet L, Wolf JP, Drouineaud V, Abdoul H, Patrat C, Denys P, Giuliano F. Prospective analysis over time of semen parameters in spinal cord-injured patients: Results of a pilot study. Andrology. 2022 Jan;10(1):120-127. doi: 10.1111/andr.13089. Epub 2021 Aug 13. PMID 34347944
- [Background] Iremashvili V, Brackett NL, Ibrahim E, Aballa TC, Lynne CM. Semen quality remains stable during the chronic phase of spinal cord injury: a longitudinal study. J Urol. 2010 Nov;184(5):2073-7. doi: 10.1016/j.juro.2010.06.112. Epub 2010 Sep 17. PMID 20850834
- [Background] Padron OF, Brackett NL, Sharma RK, Lynne CM, Thomas AJ Jr, Agarwal A. Seminal reactive oxygen species and sperm motility and morphology in men with spinal cord injury. Fertil Steril. 1997 Jun;67(6):1115-20. doi: 10.1016/s0015-0282(97)81448-3. PMID 9176453
- [Background] Brackett NL, Ibrahim E, Grotas JA, Aballa TC, Lynne CM. Higher sperm DNA damage in semen from men with spinal cord injuries compared with controls. J Androl. 2008 Jan-Feb;29(1):93-9; discussion 100-1. doi: 10.2164/jandrol.107.003574. Epub 2007 Sep 5. PMID 17804864